CLINICAL TRIAL: NCT03049683
Title: Clinical Utility of Simultaneous Recordings of Cervical and Ocular Vestibular-evoked Myogenic Potentials During Monaural Stimulation
Brief Title: Simultaneous Recordings of Cervical and Ocular Vestibular-evoked Myogenic Potentials
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chonbuk National University (Other)
Responsible Party: Principal Investigator, Sun-Young Oh, Professor, Chonbuk National University
Other Study IDs: ChonbukNU
Record Dates: First submitted 2016-12-21; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Vestibular Function Disorder
Keywords: Vestibular evoked myogenic potentials
MeSH Terms: conditions — Vestibular Diseases | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal subjects: Thirty healthy volunteers without a previous history of vertigo or neuro-otologic diseases will be enrolled in this study. The subjects will be also screened with a full history on vestibular disorders, with pure tone audiogram, and head-impulse tests to exclude the possibility of previous vestibular disorders or migraine which may cause abnormal VEMPs.
  Interventions: Other: Vestibular evoked myogenic potentials (VEMPs)
- Acute unilateral vestibular neuritis: The criteria for inclusion as a patient with vestibular neuritis involving the superior division (superior VN) included the following: (1) acute onset of vertigo, (2) the appearance of mixed horizontal and torsional nystagmus, (3) impaired horizontal semicircular canal (SCC) function on head-impulse test and a unilaterally absent or reduced caloric response (i.e., a caloric paresis score > 25%), (4) intact inferior division of vestibular nerve as evidenced by normal cVEMP and normal head-impulse test for vertical SCCs, and (5) the absence of auditory and neurologic signs. Thirty patients (aged 32-82 years; mean age, 51.7 years; 16 males) fulfilled the criteria of superior VN.
  Interventions: Other: Vestibular evoked myogenic potentials (VEMPs)

INTERVENTIONS:
Other: Vestibular evoked myogenic potentials (VEMPs) — The c- and oVEMPs will be assessed in three different sessions including conventional sequential recordings and two different simultaneous recording methods, i.e., unilateral simultaneous recording of cVEMPs and oVEMPs during monaural stimulation (Figure 1A) and bilateral simultaneous recording of each VEMP during binaural stimulation (Figure 1B).

SUMMARY:
To lower the threshold for clinical application by reducing the testing time for recording vestibular-evoked myogenic potentials (VEMPs), we evaluated whether a simultaneous recording of ocular and cervical VEMPs after unilateral or bilateral stimulation can be achieved without a loss in diagnostic sensitivity.

DETAILED DESCRIPTION:
The combined evaluation of ocular and cervical VEMPs permits the assessment of both endorgans and whole vestibular nerve function, as well as the ascending and descending vestibular pathways in the brainstem at once.

In about 30 healthy participants and 20 patients with acute unilateral vestibular neuritis, unilateral simultaneous cVEMP and oVEMP recordings in each side during monaural stimulation (air-conducted sound, 500Hz tone bursts, 100 nHL), and bilateral simultaneous recordings of each VEMP while binaural stimulation were compared to the conventional method of sequential recording each VEMPs on each side at a time.

ELIGIBILITY:
Inclusion Criteria:

1. acute onset of vertigo
2. the appearance of mixed horizontal and torsional nystagmus
3. impaired horizontal semicircular canal (SCC) function on head-impulse test and a unilaterally absent or reduced caloric response (i.e., a caloric paresis score > 25%)
4. intact inferior division of vestibular nerve as evidenced by normal cVEMP and normal head-impulse test for vertical SCCs
5. the absence of auditory and neurologic signs

Exclusion Criteria:

* a previous history of vertigo or neuro-otologic diseases

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: About thirty healthy volunteers without a previous history of vertigo or neuro-otologic diseases will be enrolled in this study. The subjects were also screened with a full history on vestibular disorders, with pure tone audiogram, and head-impulse tests to exclude the possibility of previous vestibular disorders or migraine which may cause abnormal VEMPs.
  The criteria for inclusion as a patient with vestibular neuritis involving the superior division (superior VN) will be included the following: (1) acute onset of vertigo, (2) the appearance of mixed horizontal and torsional nystagmus, (3) impaired horizontal semicircular canal (SCC) function on head-impulse test and a unilaterally absent or reduced caloric response (i.e., a caloric paresis score > 25%), (4) intact inferior division of vestibular nerve as evidenced by normal cVEMP and normal head-impulse test for vertical SCCs, and (5) the absence of auditory and neurologic signs.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Clinical utility of simultaneous recordings of cervical and ocular vestibular-evoked myogenic potentials during monaural stimulation | 6 months
  The changes in the mean time for each recording

SECONDARY OUTCOMES:
Clinical utility of simultaneous recordings of cervical and ocular vestibular-evoked myogenic potentials during monaural stimulation | 6 months
  VEMP parameters: latency
Clinical utility of simultaneous recordings of cervical and ocular vestibular-evoked myogenic potentials during monaural stimulation | 6 months
  VEMP parameters: peak-to-peak amplitude
Clinical utility of simultaneous recordings of cervical and ocular vestibular-evoked myogenic potentials during monaural stimulation | 6 months
  VEMP parameters: threshold

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh SY, Shin HJ, Boegle R, Ertl M, Eulenburg PZ, Kim JS, Dieterich M. Simultaneous recording of cervical and ocular vestibular-evoked myogenic potentials. Neurology. 2018 Jan 16;90(3):e230-e238. doi: 10.1212/WNL.0000000000004835. Epub 2017 Dec 20. PMID 29263227